CLINICAL TRIAL: NCT06258473
Title: Addressing Gaps in the Hypertension and Diabetes Care Continuum in Rural Bangladesh Through mHealth and Decentralized Primary Care: The Dinajpur Study
Brief Title: Addressing Gaps in the Hypertension and Diabetes Care Continuum in Rural Bangladesh: The Dinajpur Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BRAC University (Other)
Collaborators: Imperial College London (Other); Nanyang Technological University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-16 November-23-041
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Diabetes
Keywords: Hypertension; Diabetes; Care continumm; mHealth; Decentralized Primary Care; Rural Bangladesh
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multicomponent decentralized care (Experimental): mHealth plus decentralized primary care The multi-component intervention aims to increase access to primary care, and to improve care quality and patient retention. The intervention package includes mHealth, decentralization with task sharing, community-based care, and supportive monitoring visits
  Interventions: Combination Product: Multicomponent decentralized care; Combination Product: mHealth
- mHealth (Active Comparator): In subdistrict with mHealth intervention only, we will provide the same training on hypertension and diabetes care to physicians and nurses at NCD corner in UHC, and training to use Simple App for hypertension and diabetes management. Quarterly supervision by higher-level health administrators and medical professionals to NCD corner helps solve issues with patient management, medication supply, etc. Visits may be informed by a performance summary made available by the Simple App dashboard. Two supportive visits by the study team will be organized to help NCD Corner solve technical issues with Simple App. The healthcare providers at NCD Corner will decide how they react to the information made available by the digital tool, and similarly, the patient component will not be included. Patient pathways remain the same as usual care.
  Interventions: Combination Product: mHealth
- Usual care (No Intervention): Existing usual care provided by government primary care system including screening, treatment initiating, drug refill, and routine follow-up, at subdistrict NCD corner. Community clinics and CHWs have less involvement in NCD care provision.

INTERVENTIONS:
Combination Product: Multicomponent decentralized care — 1. Training and support on Simple app for HTN/DM management & training NCD corner clinicians on clinical guidelines and establish team-based care for Upazila level NCD corner
  2. CHCPs conduct BP/BG screening, monitoring, lifestyle counseling, dispensing of medications, follow-up overdue patients at CCs & CHCP care coordination supported by Simple app at community clinics
  3. CHWs assist in screening, counselling, referral, and follow-up for CHW at village level
  Arms: Multicomponent decentralized care
Combination Product: mHealth — Training and support on Simple app for HTN/DM patient management & training NCD corner clinicians on clinical guidelines of Upazila Health complex
  Arms: Multicomponent decentralized care; mHealth

SUMMARY:
In the present implementation study, we aim to document the experience of implementing integrated, decentralized primary care in rural Bangladesh, including components of healthcare provider training, mHealth, decentralization with task shifting, and community-based care, and to generate data on the effectiveness and cost-effectiveness of the multicomponent integrated care as compared to usual care and to mHealth intervention alone. We will also Investigate the factors that explain how the interventions influence hypertension and diabetes management and explore barriers/facilitators to delivering and sustaining intervention. We will conduct mixed-methods research to understand how the intervention influences treatment and prevention in this patient population. Particularly, we will assess lifestyle changes (i.e., smoking, dietary salt intake, physical activity, alcohol consumption), and burden for patients (e.g., waiting time, travel-related cost) at individual and community level. Qualitative data will shed light on facilitators and barriers to hypertension and diabetes prevention and control from the perspectives of patients (and their families), primary care providers, public health officials, and other stakeholders. Additionally, we will undertake a health economic evaluation of the interventions for primary care systems. A comprehensive evaluation of cost and effectiveness will be important for the models tested, providing necessary evidence for policymakers and stakeholders to scale up the interventions. We hypothesize that compared with usual care, the multicomponent decentralized primary care will improve all steps along hypertension and diabetes care continuum. On the other hand, we hypothesize that the mHealth intervention alone (Simple App) may improve BP and glycemic control compared with usual care but will have a limited impact on rates of screening, diagnosis, and treatment. We also hypothesize that the multicomponent integrated care will lead to a higher treatment success rate relative to mHealth intervention alone.

DETAILED DESCRIPTION:
Background:

Hypertension is the predominant risk factor for cardiovascular diseases (CVDs) - the leading cause of death worldwide. In 2015, 1 in 5 adult women and close to 1 in 4 adult men had elevated blood pressure. The estimated number of adults with elevated blood pressure increased from 594 million in 1975 to 1.13 billion in 2015, largely due to increases in low- and middle-income countries (LMICs).3 Globally, 10.5% adult population has diabetes, with almost half unaware of the condition they are living with. Complications of persistently elevated blood pressure and poor glycemic control, such as heart disease, stroke, chronic kidney disease, blindness, are well documented. Compared with patients with controlled blood pressure, hypertension patients without treatment and those treated but with uncontrolled blood pressure have substantially higher risk of all-cause and CVD mortality. The factors underlying the gaps in hypertension and diabetes care continuum (i.e., screening, diagnosis, treatment, control) are complex and multifactorial, reflecting the vulnerabilities at individual, community, and healthcare system levels in LMICs.Few studies have examined the strategy to address shortage of healthcare human resources and NCD care accessibility through decentralization with task shifting (or task sharing), which has been shown a viable strategy to rapidly scale-up antiretroviral therapy for HIV/AIDS care in resource-limited settings. Like many other LMICs, Bangladesh is experiencing rapid demographic and epidemiologic transitions. In the recent years, NCD replaced infectious disease and maternal and neonatal conditions as the leading cause of death, accounting for 71% of all deaths in Bangladesh. An estimated 27.4% of Bangladeshi adults have hypertension and 9.8% have diabetes. According to 2017-2018 Bangladesh Demographic and Health Survey, only 36.7% of Bangladeshi adults with hypertension were aware that they had hypertension, and only 31.1% were on treatment and 12.7% had blood pressure controlled. The awareness, treatment, and control rates for diabetes were estimated to be 30.9%, 28.2%, and 26.5%, respectively. Tobacco use, insufficient fruit/vegetable intake, overweight/obese, are highly prevalent. Over the past decade, the Government of Bangladesh has promoted improved NCD care through national multisectoral actions, most notably through the establishment of dedicated noncommunicable disease facilities ("NCD Corners") at subdistrict hospitals since 2011. These NCD Corners were designed to provide preventive and clinical care for common NCDs. Despite the initiative, NCD corners remained nascent due to a lack of specific guidelines, trained workforce, appropriate medicines and supplies, adequate laboratory facilities, and poor record-keeping and reporting.

In the present study, we aim to document the experience of implementing a multicomponent, decentralized primary care in rural Bangladesh, including components of healthcare provider training, mHealth, decentralization with task shifting, and community-based care, and to generate data on the effectiveness and cost-effectiveness of the multicomponent integrated care as compared to usual care and to mHealth intervention alone.

Study design

This is a type 2 effectiveness-implementation hybrid study with a dual focus on testing of effectiveness of interventions and implementation strategies.41 A three-arm mixed-methods quasi-experimental design will be used to achieve the aims specified before. Two intervention subdistricts (i.e., mHealth only and mHealth plus task sharing, decentralization, and community-based care) and one reference subdistrict from Dinajpur district, Rangpur division in Northern Bangladesh (Figure 1) will be selected to implement the study. While the key outcomes will be evaluated with community-based repeated cross-sectional surveys with independent samples, we will also make use of facility-based prospective cohort data to supplement community-based surveys. We will employ a mixed methods approach to generate rich data on changes in primary and secondary outcomes, and quantitative and qualitative data for process evaluation. The project duration is 36 months.

Specific objectives and hypothesis of the study

SA1: Document the experience of implementing a multicomponent decentralized care in public primary care system for hypertension and diabetes and evaluate the effectiveness of the package compared with usual care and mHealth intervention alone. The findings will not only shed light on the effectiveness of the interventions on treatment outcomes, but will also informing approaches to improve screening, diagnosis, and management of these conditions. Among the first, we expect to provide data on the role of decentralization for expanding NCD care in resource limited settings.

SA2: Investigate the factors that explain how the interventions influences hypertension and diabetes management and explore barriers/facilitators to deliver and sustaining intervention. We will conduct mixed methods research to understand how the intervention influences treatment and prevention in this patient population. Particularly, we will assess changes in lifestyle (i.e., smoking, dietary salt intake, physical activity, alcohol consumption), burden for patients (e.g., waiting time, travel-related cost) at individual and community level. Qualitative data will shed light on facilitators and barriers to hypertension and diabetes prevention and control from perspectives of patients (and their families), primary care providers, and public health officials, and other stakeholders.

SA3: Undertake a health economic evaluation of the interventions for primary care systems. A comprehensive evaluation of cost and effectiveness will be important for the models tested, providing necessary evidence for policy makes and stakeholders to scale up the interventions.

We hypothesize that compared with usual care, the multicomponent decentralized primary care will improve all steps along the hypertension and diabetes care continuum. On the other hand, we hypothesize that the mHealth intervention alone (Simple App) may improve BP and glycemic control compared with usual care but will have limited impact on rates of screening, diagnosis, and treatment. We also hypothesize that the multicomponent integrated care will lead to higher treatment success rate relative to mHealth intervention alone.

Study population and settings:

In rural Bangladesh, a subdistrict (Upazila) is the second lowest tier of administration, while union is the lowest rural administrative unit, and each union is made up of nine wards (usually one village is designated as a ward). The primary healthcare system in rural areas consist of a subdistrict level hospital (Upazila Health Complexes), union health (sub)centers, and community clinics which cover 2 to 4 villages. A Upazila Health Complex lies at the top of the primary care system. It is typically a 50-bed hospital, serving a population of a few hundred thousand.

Community clinics are at the lowest level of the healthcare facility hierarchy. With two rooms and drinking-water and lavatory facilities under a covered waiting area, community clinics were designed to be accessible for more than 80% of rural population within less than 30-minute walking distance.42 Community clinics are staffed by a Community Health Care Provider (CHCP), who usually receive 4-month medical training.

Interventions

Built upon assessment of barriers to hypertension and diabetes management at patient, provider, and health system levels and previous interventional studies, a multicomponent intervention package was designed to increase access to primary care, and to improve care quality and patient retention. The intervention package includes mHealth, decentralization with task sharing, community-based care, and supportive monitoring visits. The effectiveness of the intervention package is compared with mHealth only intervention and usual care.

Description of the interventions Multicomponent decentralized care

It will include both government model and mHealth for patient management and some other components like supportive supervisions. In line with Bangladesh government's recommendation, Simple App will be used by primary care facilities for coordinated NCD management. The Simple App was developed and is actively maintained by Resolve to Save Lives (more details about the app can be found from the website https://www.simple.org). The app was designed to tackle two major factors contribute to blood pressure and glycemic control among treated patients with hypertension and diabetes, namely timely titration and adherence with therapy. To accommodate the context of busy primary care facilities, data collection is limited to a few key variables such as prescription, follow-up visit, and changes in blood pressure and blood glucose. Using unique patient ID, the app allows seamless transferring of electronic health records among primary care facilities and thus ensure continuity of the process.

Engaging community health workers in NCD care: Integrating hypertension and diabetes care into the community by training CHWs to provide screening, counselling, and follow-up has been shown to improve hypertension and diabetes care management in many LMICs, including countries from South Asia. In line with previous studies, we will enlist CHWs in case finding, counselling, referral, and follow-up. Existing CHWs will be trained and provided with necessary equipment and health education materials and tools to carry out these tasks. Initial training will cover topics including basics of hypertension and diabetes, lifestyle risk factors counselling, patient self-management, and collaboration with CHCPs. A refresher training will be done at 6 months of implementation. CHWs will not be compensated for the activities performed to be consistent with Bangladesh government's plan considering scalability.

Supportive monitoring and supervision: Quarterly supervision by higher level health administrators and medical professionals will be organized to NCD corner to help solve issues with patient managements, medication supply etc. Visits may be informed by performance summary made available by Simple App dashboard. Similarly, quarterly supervision to CCs by NCD corner medical staff and subdistrict health officials will be done. Supportive visits by study team will be organized to help NCD corners and CCs solve technical issues with Simple App.

mHealth only

In subdistrict with mHealth intervention only, training and support to use Simple App for hypertension and diabetes management will be provided. The healthcare providers at NCD corner will decide how they react to the information made available by the digital tool, and similarly the patient component will not be included. Patient pathways remain the same as usual care.

Usual care

Existing usual care provided by government primary care system including screening, treatment initiating, drug refill, and routine follow-up, at subdistrict NCD corner. Community clinics and CHWs have less involvement in NCD care provision.

ELIGIBILITY:
Inclusion Criteria:

* All participants aged 40 or above
* With hypertension and diabetes
* Residents of specific study areas
* Willing to participate

Exclusion Criteria:

* Adults aged less than 40 years
* Children
* Pregnant women
* Severely ill
* Having severe disabilities both physical and mental)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6750 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hypertension and Diabetes control | 2 years and 9 months
  The primary outcome will be the proportion of patients treated for NCDs who achieved or maintained disease-specific controlled status, according to national or WHO PEN protocols. Hypertension is considered controlled if SBP<140 mmHg and DBP<90 mmHg for most patients, and if SBP<130 mmHg and DBP<80 mmHg for patients who have comorbidities (diabetes, heart disease, stroke, chronic kidney disease) or having 10-year CVD risk ≥ 30%. Goal for glycemic control is fasting plasma glucose 4.4-7.2 mmol/L, or random plasma glucose <11.1 mmol/L. The effectiveness will be assessed primarily using repeated independent community-based surveys.

SECONDARY OUTCOMES:
Hypertension and diabetes care cascade | 2 years and 9 months
  Secondary outcomes include hypertension and diabetes care cascade (i.e. % of patients aware of their condition, % of diagnosed patients on treatment), smoking cessation among HTN/DM patients, and meeting recommended physical activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Malay K Mridha, PhD, Principal Investigator — BRAC University - School of Public Health; John C Chambers, PhD, Principal Investigator — Imperial College London
Locations (1):
- BRAC James P Grant School of Public Health, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun H, Saeedi P, Karuranga S, Pinkepank M, Ogurtsova K, Duncan BB, Stein C, Basit A, Chan JCN, Mbanya JC, Pavkov ME, Ramachandaran A, Wild SH, James S, Herman WH, Zhang P, Bommer C, Kuo S, Boyko EJ, Magliano DJ. IDF Diabetes Atlas: Global, regional and country-level diabetes prevalence estimates for 2021 and projections for 2045. Diabetes Res Clin Pract. 2022 Jan;183:109119. doi: 10.1016/j.diabres.2021.109119. Epub 2021 Dec 6. PMID 34879977
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in blood pressure from 1975 to 2015: a pooled analysis of 1479 population-based measurement studies with 19.1 million participants. Lancet. 2017 Jan 7;389(10064):37-55. doi: 10.1016/S0140-6736(16)31919-5. Epub 2016 Nov 16. PMID 27863813
- [Background] Gu Q, Dillon CF, Burt VL, Gillum RF. Association of hypertension treatment and control with all-cause and cardiovascular disease mortality among US adults with hypertension. Am J Hypertens. 2010 Jan;23(1):38-45. doi: 10.1038/ajh.2009.191. Epub 2009 Oct 22. PMID 19851295
- [Background] Gu Q, Burt VL, Paulose-Ram R, Yoon S, Gillum RF. High blood pressure and cardiovascular disease mortality risk among U.S. adults: the third National Health and Nutrition Examination Survey mortality follow-up study. Ann Epidemiol. 2008 Apr;18(4):302-9. doi: 10.1016/j.annepidem.2007.11.013. Epub 2008 Feb 8. PMID 18261929
- [Background] Manne-Goehler J, Geldsetzer P, Agoudavi K, Andall-Brereton G, Aryal KK, Bicaba BW, Bovet P, Brian G, Dorobantu M, Gathecha G, Singh Gurung M, Guwatudde D, Msaidie M, Houehanou C, Houinato D, Jorgensen JMA, Kagaruki GB, Karki KB, Labadarios D, Martins JS, Mayige MT, McClure RW, Mwalim O, Mwangi JK, Norov B, Quesnel-Crooks S, Silver BK, Sturua L, Tsabedze L, Wesseh CS, Stokes A, Marcus M, Ebert C, Davies JI, Vollmer S, Atun R, Barnighausen TW, Jaacks LM. Health system performance for people with diabetes in 28 low- and middle-income countries: A cross-sectional study of nationally representative surveys. PLoS Med. 2019 Mar 1;16(3):e1002751. doi: 10.1371/journal.pmed.1002751. eCollection 2019 Mar. PMID 30822339
- [Background] Geldsetzer P, Manne-Goehler J, Marcus ME, Ebert C, Zhumadilov Z, Wesseh CS, Tsabedze L, Supiyev A, Sturua L, Bahendeka SK, Sibai AM, Quesnel-Crooks S, Norov B, Mwangi KJ, Mwalim O, Wong-McClure R, Mayige MT, Martins JS, Lunet N, Labadarios D, Karki KB, Kagaruki GB, Jorgensen JMA, Hwalla NC, Houinato D, Houehanou C, Msaidie M, Guwatudde D, Gurung MS, Gathecha G, Dorobantu M, Damasceno A, Bovet P, Bicaba BW, Aryal KK, Andall-Brereton G, Agoudavi K, Stokes A, Davies JI, Barnighausen T, Atun R, Vollmer S, Jaacks LM. The state of hypertension care in 44 low-income and middle-income countries: a cross-sectional study of nationally representative individual-level data from 1.1 million adults. Lancet. 2019 Aug 24;394(10199):652-662. doi: 10.1016/S0140-6736(19)30955-9. Epub 2019 Jul 18. PMID 31327566
- [Background] Zhou B, Perel P, Mensah GA, Ezzati M. Global epidemiology, health burden and effective interventions for elevated blood pressure and hypertension. Nat Rev Cardiol. 2021 Nov;18(11):785-802. doi: 10.1038/s41569-021-00559-8. Epub 2021 May 28. PMID 34050340
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Long-term and recent trends in hypertension awareness, treatment, and control in 12 high-income countries: an analysis of 123 nationally representative surveys. Lancet. 2019 Aug 24;394(10199):639-651. doi: 10.1016/S0140-6736(19)31145-6. Epub 2019 Jul 18. PMID 31327564
- [Background] Bodenheimer T, Wagner EH, Grumbach K. Improving primary care for patients with chronic illness: the chronic care model, Part 2. JAMA. 2002 Oct 16;288(15):1909-14. doi: 10.1001/jama.288.15.1909. PMID 12377092
- [Background] Kabir A, Karim MN, Islam RM, Romero L, Billah B. Health system readiness for non-communicable diseases at the primary care level: a systematic review. BMJ Open. 2022 Feb 9;12(2):e060387. doi: 10.1136/bmjopen-2021-060387. PMID 35140165
- [Background] Kruk ME, Nigenda G, Knaul FM. Redesigning primary care to tackle the global epidemic of noncommunicable disease. Am J Public Health. 2015 Mar;105(3):431-7. doi: 10.2105/AJPH.2014.302392. Epub 2015 Jan 20. PMID 25602898
- [Background] Kruk ME, Gage AD, Arsenault C, Jordan K, Leslie HH, Roder-DeWan S, Adeyi O, Barker P, Daelmans B, Doubova SV, English M, Garcia-Elorrio E, Guanais F, Gureje O, Hirschhorn LR, Jiang L, Kelley E, Lemango ET, Liljestrand J, Malata A, Marchant T, Matsoso MP, Meara JG, Mohanan M, Ndiaye Y, Norheim OF, Reddy KS, Rowe AK, Salomon JA, Thapa G, Twum-Danso NAY, Pate M. High-quality health systems in the Sustainable Development Goals era: time for a revolution. Lancet Glob Health. 2018 Nov;6(11):e1196-e1252. doi: 10.1016/S2214-109X(18)30386-3. Epub 2018 Sep 5. No abstract available. PMID 30196093
- [Background] Frenk J, Chen L, Bhutta ZA, Cohen J, Crisp N, Evans T, Fineberg H, Garcia P, Ke Y, Kelley P, Kistnasamy B, Meleis A, Naylor D, Pablos-Mendez A, Reddy S, Scrimshaw S, Sepulveda J, Serwadda D, Zurayk H. Health professionals for a new century: transforming education to strengthen health systems in an interdependent world. Lancet. 2010 Dec 4;376(9756):1923-58. doi: 10.1016/S0140-6736(10)61854-5. Epub 2010 Nov 26. No abstract available. PMID 21112623
- [Background] Chowdhury HA, Paromita P, Mayaboti CA, Rakhshanda S, Rahman FN, Abedin M, Rahman AKMF, Mashreky SR. Assessing service availability and readiness of healthcare facilities to manage diabetes mellitus in Bangladesh: Findings from a nationwide survey. PLoS One. 2022 Feb 16;17(2):e0263259. doi: 10.1371/journal.pone.0263259. eCollection 2022. PMID 35171912
- [Background] Islam K, Huque R, Saif-Ur-Rahman KM, Ehtesham Kabir ANM, Enayet Hussain AHM. Implementation status of non-communicable disease control program at primary health care level in Bangladesh: Findings from a qualitative research. Public Health Pract (Oxf). 2022 May 10;3:100271. doi: 10.1016/j.puhip.2022.100271. eCollection 2022 Jun. PMID 36101774
- [Background] Correia JC, Lachat S, Lagger G, Chappuis F, Golay A, Beran D; COHESION Project. Interventions targeting hypertension and diabetes mellitus at community and primary healthcare level in low- and middle-income countries:a scoping review. BMC Public Health. 2019 Nov 21;19(1):1542. doi: 10.1186/s12889-019-7842-6. PMID 31752801
- [Background] Ye J, Orji IA, Baldridge AS, Ojo TM, Shedul G, Ugwuneji EN, Egenti NB, Aluka-Omitiran K, Okoli RCB, Eze H, Nwankwo A, Hirschhorn LR, Chopra A, Ale BM, Shedul GL, Tripathi P, Kandula NR, Huffman MD, Ojji DB; Hypertension Treatment in Nigeria Program Investigators. Characteristics and Patterns of Retention in Hypertension Care in Primary Care Settings From the Hypertension Treatment in Nigeria Program. JAMA Netw Open. 2022 Sep 1;5(9):e2230025. doi: 10.1001/jamanetworkopen.2022.30025. PMID 36066896
- [Background] Labhardt ND, Balo JR, Ndam M, Grimm JJ, Manga E. Task shifting to non-physician clinicians for integrated management of hypertension and diabetes in rural Cameroon: a programme assessment at two years. BMC Health Serv Res. 2010 Dec 14;10:339. doi: 10.1186/1472-6963-10-339. PMID 21144064
- [Background] Deo S, Singh P. Community health worker-led, technology-enabled private sector intervention for diabetes and hypertension management among urban poor: a retrospective cohort study from large Indian metropolitan city. BMJ Open. 2021 Aug 12;11(8):e045246. doi: 10.1136/bmjopen-2020-045246. PMID 34385229
- [Background] Labrique AB, Wadhwani C, Williams KA, Lamptey P, Hesp C, Luk R, Aerts A. Best practices in scaling digital health in low and middle income countries. Global Health. 2018 Nov 3;14(1):103. doi: 10.1186/s12992-018-0424-z. PMID 30390686
- [Background] Anchala R, Kaptoge S, Pant H, Di Angelantonio E, Franco OH, Prabhakaran D. Evaluation of effectiveness and cost-effectiveness of a clinical decision support system in managing hypertension in resource constrained primary health care settings: results from a cluster randomized trial. J Am Heart Assoc. 2015 Jan 5;4(1):e001213. doi: 10.1161/JAHA.114.001213. PMID 25559011
- [Background] Prabhakaran D, Jha D, Prieto-Merino D, Roy A, Singh K, Ajay VS, Jindal D, Gupta P, Kondal D, Goenka S, Jacob P, Singh R, Kumar BGP, Perel P, Tandon N, Patel V; Members of the Research Steering Committee,Investigators,Members of the Data Safety and Monitoring Board. Effectiveness of an mHealth-Based Electronic Decision Support System for Integrated Management of Chronic Conditions in Primary Care: The mWellcare Cluster-Randomized Controlled Trial. Circulation. 2019 Jan 15;139(3):380-391. doi: 10.1161/CIRCULATIONAHA.118.038192. Epub 2018 Nov 10. PMID 30586732
- [Background] Kumar A, Schwarz D, Acharya B, Agrawal P, Aryal A, Choudhury N, Citrin D, Dangal B, Deukmedjian G, Dhimal M, Dhungana S, Gauchan B, Gupta T, Halliday S, Jha D, Kalaunee SP, Karmacharya B, Kishore S, Koirala B, Kunwar L, Mahar R, Maru S, Mehanni S, Nirola I, Pandey S, Pant B, Pathak M, Poudel S, Rajbhandari I, Raut A, Rimal P, Schwarz R, Shrestha A, Thapa A, Thapa P, Thapa R, Wong L, Maru D. Designing and implementing an integrated non-communicable disease primary care intervention in rural Nepal. BMJ Glob Health. 2019 Apr 29;4(2):e001343. doi: 10.1136/bmjgh-2018-001343. eCollection 2019. PMID 31139453
- [Background] He J, Irazola V, Mills KT, Poggio R, Beratarrechea A, Dolan J, Chen CS, Gibbons L, Krousel-Wood M, Bazzano LA, Nejamis A, Gulayin P, Santero M, Augustovski F, Chen J, Rubinstein A; HCPIA Investigators. Effect of a Community Health Worker-Led Multicomponent Intervention on Blood Pressure Control in Low-Income Patients in Argentina: A Randomized Clinical Trial. JAMA. 2017 Sep 19;318(11):1016-1025. doi: 10.1001/jama.2017.11358. PMID 28975305
- [Background] Jafar TH, Gandhi M, de Silva HA, Jehan I, Naheed A, Finkelstein EA, Turner EL, Morisky D, Kasturiratne A, Khan AH, Clemens JD, Ebrahim S, Assam PN, Feng L; COBRA-BPS Study Group. A Community-Based Intervention for Managing Hypertension in Rural South Asia. N Engl J Med. 2020 Feb 20;382(8):717-726. doi: 10.1056/NEJMoa1911965. PMID 32074419
- [Background] Schwalm JD, McCready T, Lopez-Jaramillo P, Yusoff K, Attaran A, Lamelas P, Camacho PA, Majid F, Bangdiwala SI, Thabane L, Islam S, McKee M, Yusuf S. A community-based comprehensive intervention to reduce cardiovascular risk in hypertension (HOPE 4): a cluster-randomised controlled trial. Lancet. 2019 Oct 5;394(10205):1231-1242. doi: 10.1016/S0140-6736(19)31949-X. Epub 2019 Sep 2. PMID 31488369
- [Background] Brennan AT, Long L, Maskew M, Sanne I, Jaffray I, MacPhail P, Fox MP. Outcomes of stable HIV-positive patients down-referred from a doctor-managed antiretroviral therapy clinic to a nurse-managed primary health clinic for monitoring and treatment. AIDS. 2011 Oct 23;25(16):2027-36. doi: 10.1097/QAD.0b013e32834b6480. PMID 21997488
- [Background] Sanne I, Orrell C, Fox MP, Conradie F, Ive P, Zeinecker J, Cornell M, Heiberg C, Ingram C, Panchia R, Rassool M, Gonin R, Stevens W, Truter H, Dehlinger M, van der Horst C, McIntyre J, Wood R; CIPRA-SA Study Team. Nurse versus doctor management of HIV-infected patients receiving antiretroviral therapy (CIPRA-SA): a randomised non-inferiority trial. Lancet. 2010 Jul 3;376(9734):33-40. doi: 10.1016/S0140-6736(10)60894-X. PMID 20557927
- [Background] Lehmann U, Van Damme W, Barten F, Sanders D. Task shifting: the answer to the human resources crisis in Africa? Hum Resour Health. 2009 Jun 21;7:49. doi: 10.1186/1478-4491-7-49. PMID 19545398
- [Background] Kredo T, Ford N, Adeniyi FB, Garner P. Decentralising HIV treatment in lower- and middle-income countries. Cochrane Database Syst Rev. 2013 Jun 27;2013(6):CD009987. doi: 10.1002/14651858.CD009987.pub2. PMID 23807693
- [Background] Kaur P, Kunwar A, Sharma M, Durgad K, Gupta S; India Hypertension Control Initiative collaboration; Bhargava B. The India Hypertension Control Initiative-early outcomes in 26 districts across five states of India, 2018-2020. J Hum Hypertens. 2023 Jul;37(7):560-567. doi: 10.1038/s41371-022-00742-5. Epub 2022 Aug 9. PMID 35945426
- [Background] Patel SA, Sharma H, Mohan S, Weber MB, Jindal D, Jarhyan P, Gupta P, Sharma R, Ali M, Ali MK, Narayan KMV, Prabhakaran D, Gupta Y, Roy A, Tandon N. The Integrated Tracking, Referral, and Electronic Decision Support, and Care Coordination (I-TREC) program: scalable strategies for the management of hypertension and diabetes within the government healthcare system of India. BMC Health Serv Res. 2020 Nov 9;20(1):1022. doi: 10.1186/s12913-020-05851-w. PMID 33168004
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Khan N, Oldroyd JC, Hossain MB, Islam RM. Awareness, Treatment, and Control of Diabetes in Bangladesh: Evidence from the Bangladesh Demographic and Health Survey 2017/18. Int J Clin Pract. 2022 Apr 22;2022:8349160. doi: 10.1155/2022/8349160. eCollection 2022. PMID 35685557
- [Background] Khan MN, Oldroyd JC, Chowdhury EK, Hossain MB, Rana J, Renzetti S, Islam RM. Prevalence, awareness, treatment, and control of hypertension in Bangladesh: Findings from National Demographic and Health Survey, 2017-2018. J Clin Hypertens (Greenwich). 2021 Oct;23(10):1830-1842. doi: 10.1111/jch.14363. Epub 2021 Sep 7. PMID 34492733
- [Background] Riaz BK, Islam MZ, Islam ANMS, Zaman MM, Hossain MA, Rahman MM, Khanam F, Amin KMB, Noor IN. Risk factors for non-communicable diseases in Bangladesh: findings of the population-based cross-sectional national survey 2018. BMJ Open. 2020 Nov 27;10(11):e041334. doi: 10.1136/bmjopen-2020-041334. PMID 33247026
- [Background] Burka D, Gupta R, Moran AE, Cohn J, Choudhury SR, Cheadle T, Mullick R, Frieden TR. Keep it simple: designing a user-centred digital information system to support chronic disease management in low/middle-income countries. BMJ Health Care Inform. 2023 Jan;30(1):e100641. doi: 10.1136/bmjhci-2022-100641. PMID 36639189
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Chowdhury AM, Bhuiya A, Chowdhury ME, Rasheed S, Hussain Z, Chen LC. The Bangladesh paradox: exceptional health achievement despite economic poverty. Lancet. 2013 Nov 23;382(9906):1734-45. doi: 10.1016/S0140-6736(13)62148-0. Epub 2013 Nov 21. PMID 24268002
- [Background] Schwalm JD, McKee M, Huffman MD, Yusuf S. Resource Effective Strategies to Prevent and Treat Cardiovascular Disease. Circulation. 2016 Feb 23;133(8):742-55. doi: 10.1161/CIRCULATIONAHA.115.008721. PMID 26903017
- [Background] Naheed A, Haldane V, Jafar TH, Chakma N, Legido-Quigley H. Patient pathways and perceptions of hypertension treatment, management, and control in rural Bangladesh: a qualitative study. Patient Prefer Adherence. 2018 Aug 14;12:1437-1449. doi: 10.2147/PPA.S163385. eCollection 2018. PMID 30147302
- [Background] Legido-Quigley H, Naheed A, de Silva HA, Jehan I, Haldane V, Cobb B, Tavajoh S, Chakma N, Kasturiratne A, Siddiqui S, Jafar TH; for COBRA-BPS Study group. Patients' experiences on accessing health care services for management of hypertension in rural Bangladesh, Pakistan and Sri Lanka: A qualitative study. PLoS One. 2019 Jan 25;14(1):e0211100. doi: 10.1371/journal.pone.0211100. eCollection 2019. PMID 30682093
- [Background] Nam S, Chesla C, Stotts NA, Kroon L, Janson SL. Barriers to diabetes management: patient and provider factors. Diabetes Res Clin Pract. 2011 Jul;93(1):1-9. doi: 10.1016/j.diabres.2011.02.002. Epub 2011 Mar 5. PMID 21382643
- [Background] Burnier M, Egan BM. Adherence in Hypertension. Circ Res. 2019 Mar 29;124(7):1124-1140. doi: 10.1161/CIRCRESAHA.118.313220. PMID 30920917
- [Background] Abrahams-Gessel S, Denman CA, Montano CM, Gaziano TA, Levitt N, Rivera-Andrade A, Carrasco DM, Zulu J, Khanam MA, Puoane T. The training and fieldwork experiences of community health workers conducting population-based, noninvasive screening for CVD in LMIC. Glob Heart. 2015 Mar;10(1):45-54. doi: 10.1016/j.gheart.2014.12.008. PMID 25754566
- [Background] Alaofe H, Asaolu I, Ehiri J, Moretz H, Asuzu C, Balogun M, Abosede O, Ehiri J. Community Health Workers in Diabetes Prevention and Management in Developing Countries. Ann Glob Health. 2017 May-Aug;83(3-4):661-675. doi: 10.1016/j.aogh.2017.10.009. Epub 2017 Nov 22. PMID 29221543
- [Background] Anand TN, Joseph LM, Geetha AV, Prabhakaran D, Jeemon P. Task sharing with non-physician health-care workers for management of blood pressure in low-income and middle-income countries: a systematic review and meta-analysis. Lancet Glob Health. 2019 Jun;7(6):e761-e771. doi: 10.1016/S2214-109X(19)30077-4. PMID 31097278
- [Background] Gaziano TA, Abrahams-Gessel S, Denman CA, Montano CM, Khanam M, Puoane T, Levitt NS. An assessment of community health workers' ability to screen for cardiovascular disease risk with a simple, non-invasive risk assessment instrument in Bangladesh, Guatemala, Mexico, and South Africa: an observational study. Lancet Glob Health. 2015 Sep;3(9):e556-63. doi: 10.1016/S2214-109X(15)00143-6. Epub 2015 Jul 14. PMID 26187361
- [Background] Schwarz D, Dhungana S, Kumar A, Acharya B, Agrawal P, Aryal A, Baum A, Choudhury N, Citrin D, Dangal B, Dhimal M, Gauchan B, Gupta T, Halliday S, Karmacharya B, Kishore S, Koirala B, Kshatriya U, Levine E, Maru S, Rimal P, Sapkota S, Schwarz R, Shrestha A, Thapa A, Maru D. An integrated intervention for chronic care management in rural Nepal: protocol of a type 2 hybrid effectiveness-implementation study. Trials. 2020 Jan 29;21(1):119. doi: 10.1186/s13063-020-4063-3. PMID 31996250
- [Background] Song P, Gupta A, Goon IY, Hasan M, Mahmood S, Pradeepa R, Siddiqui S, Frost GS, Kusuma D, Miraldo M, Sassi F, Wareham NJ, Ahmed S, Anjana RM, Brage S, Forouhi NG, Jha S, Kasturiratne A, Katulanda P, Khawaja KI, Loh M, Mridha MK, Wickremasinghe AR, Kooner JS, Chambers JC; South Asia Biobank. Remaining authors are listed at the end of the article. Data Resource Profile: Understanding the patterns and determinants of health in South Asians-the South Asia Biobank. Int J Epidemiol. 2021 Jul 9;50(3):717-718e. doi: 10.1093/ije/dyab029. No abstract available. PMID 34143882
- [Background] Gandhi M, Assam PN, Turner EL, Morisky DE, Chan E, Jafar TH; COBRA-BPS Study Group. Statistical analysis plan for the control of blood pressure and risk attenuation-rural Bangladesh, Pakistan, Sri Lanka (COBRA-BPS) trial: a cluster randomized trial for a multicomponent intervention versus usual care in hypertensive patients. Trials. 2018 Nov 29;19(1):658. doi: 10.1186/s13063-018-3022-8. PMID 30486858
- [Background] Xie W, Paul RR, Goon IY, Anan A, Rahim A, Hossain MM, Hersch F, Oldenburg B, Chambers J, Mridha MK. Enhancing care quality and accessibility through digital technology-supported decentralisation of hypertension and diabetes management: a proof-of-concept study in rural Bangladesh. BMJ Open. 2023 Nov 19;13(11):e073743. doi: 10.1136/bmjopen-2023-073743. PMID 37984955
- [Background] Campbell MJ, Julious SA, Altman DG. Estimating sample sizes for binary, ordered categorical, and continuous outcomes in two group comparisons. BMJ. 1995 Oct 28;311(7013):1145-8. doi: 10.1136/bmj.311.7013.1145. PMID 7580713
- [Background] Lipsitch M, Tchetgen Tchetgen E, Cohen T. Negative controls: a tool for detecting confounding and bias in observational studies. Epidemiology. 2010 May;21(3):383-8. doi: 10.1097/EDE.0b013e3181d61eeb. PMID 20335814
- [Background] Zou GY, Donner A. Extension of the modified Poisson regression model to prospective studies with correlated binary data. Stat Methods Med Res. 2013 Dec;22(6):661-70. doi: 10.1177/0962280211427759. Epub 2011 Nov 8. PMID 22072596
- [Background] Yelland LN, Salter AB, Ryan P. Performance of the modified Poisson regression approach for estimating relative risks from clustered prospective data. Am J Epidemiol. 2011 Oct 15;174(8):984-92. doi: 10.1093/aje/kwr183. Epub 2011 Aug 12. PMID 21841157
- [Background] Xu X, Lazar CM, Ruger JP. Micro-costing in health and medicine: a critical appraisal. Health Econ Rev. 2021 Jan 6;11(1):1. doi: 10.1186/s13561-020-00298-5. PMID 33404857
- [Background] Sanders GD, Neumann PJ, Basu A, Brock DW, Feeny D, Krahn M, Kuntz KM, Meltzer DO, Owens DK, Prosser LA, Salomon JA, Sculpher MJ, Trikalinos TA, Russell LB, Siegel JE, Ganiats TG. Recommendations for Conduct, Methodological Practices, and Reporting of Cost-effectiveness Analyses: Second Panel on Cost-Effectiveness in Health and Medicine. JAMA. 2016 Sep 13;316(10):1093-103. doi: 10.1001/jama.2016.12195. PMID 27623463
- [Background] Oti SO, van de Vijver S, Gomez GB, Agyemang C, Egondi T, Kyobutungi C, Stronks K. Outcomes and costs of implementing a community-based intervention for hypertension in an urban slum in Kenya. Bull World Health Organ. 2016 Jul 1;94(7):501-9. doi: 10.2471/BLT.15.156513. Epub 2016 Apr 26. PMID 27429489